CLINICAL TRIAL: NCT05094011
Title: A Phase I Open-Label Dose-Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of Autologous MitoCell (Adipose-Derived Mesenchymal Stem Cells) Transplantation in Subjects With Idiopathic Parkinson's Disease
Brief Title: Evaluating Safety, Tolerability, and Efficacy of Autologous MitoCell Transplantation in Subjects With Idiopathic Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiwan Mitochondrion Applied Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MITOCELL-01
Record Dates: First submitted 2021-07-20; First posted 2021-10-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study plans to enroll approximately 4 subjects to obtain 3 evaluable subjects successfully receiving 3×10^7 cells/hemisphere (total 6×10^7 cells, Cohort 1) and approximately 8 subjects to obtain 6 evaluable subjects for 1×10^8 cells/hemisphere (total 2×10^8 cells, Cohort 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): Autologous MitoCell Transplantation in Subjects with Idiopathic Parkinson's Disease
  Interventions: Biological: Aadipose-Derived Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Aadipose-Derived Mesenchymal Stem Cells — Stereotactic intrastriatal implantation of 3×10^7 per hemisphere (total 6×10^7 cells) or 1×10^8 per hemisphere (total 2×10^8 cells) autologous TM01-treated adipose-derived mesenchymal stem cells (MitoCell).
  Other Names: MitoCell

SUMMARY:
Primary Objective: To assess the safety profile of autologous MitoCell administered to subjects with idiopathic Parkinson's disease (PD)

Secondary Objective: To explore the efficacy and safety of MitoCell given as the recommended dose by stereotactic intrastriatal implantation

DETAILED DESCRIPTION:
MitoCell is an autologous stem cell product that cultures with the company's unique patented medium. The mechanism of action of MitoCell is to improve the brain microenvironment in neurodegenerative disease. MitoCell which like mesenchymal stem cells modulate the immune response, and secrete more BDNF and SDF-1 neurotrophic factors than regular stem cell products.Therefore, MitoCell can protect and repair damaged dopamine neurons (DA) and stimulate DA regeneration.This project is a phase I open-label dose-escalation study to evaluate the safety, tolerability, and efficacy of autologous MitoCell intracranial transplantation in subjects with idiopathic Parkinson's disease which rating from stage 3 ~ 4 of modified Hoehn & Yahr staging.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Aged 45 to 70 years old (inclusive) at Screening
* Idiopathic Parkinson's disease patients who meet the diagnostic criteria of the "Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease"
* With at least 5 years since the diagnosis of Parkinson's disease
* With responsiveness to levodopa or dopa agonist. This is defined as improvement between ''Off'' and ''On'' MDS-UPDRS by at least 33% of the Motor MDS-UPDRS
* Idiopathic Parkinson's disease of Stage 3 ~ 4 of modified Hoehn & Yahr staging during ''ON'' time
* Stable Parkinsonian medications for at least 2 months prior to the Screening Visit
* MRI not showing gross atrophy or any brain pathology other than PD
* Mini-Mental State Examination (MMSE) ≧ 24
* With score of the Beck Depression Inventory (BDI-II) < 29 and Hamilton Rating Scale for Depression (HAM-D-17) < 25

Exclusion Criteria:

* Atypical or secondary Parkinsonism
* With neurodegenerative disorders other than PD
* Unable to receive MRI or PET scanning
* With any concomitant disorder that would contraindicate coagulation, general anesthesia, or stereotactic neurosurgery
* Received any other investigational agent within 4 weeks prior to Screening
* History of intracranial surgeries or implantation of a device for Parkinson's disease 2 years prior to Screening
* Major surgery within the previous 6 months at Screening
* Significant cardiovascular disease, including:

  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Uncontrolled hypertension: Blood pressure >140/90 mmHg
  * History of serious ventricular arrhythmia
* Malignancy within 2 years prior to Screening
* Any diagnosis of autoimmune disease or immune compromised state and requiring systemic steroid or immunosuppressive treatment
* Any other severe systemic disorder, including history of schizophrenia or other psychotic disorders, stroke, seizure, traumatic brain injury, or central nervous system infection, which judged by the investigator that entering the trial may be detrimental to the subject
* Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent and perform all study assessments
* Positive in any of the following regulatory authority-licensed screening tests:

  * HIV antigen/antibody combo test
  * Anti-HCV test
  * Hepatitis B surface antigen (HBsAg) test
  * Rapid plasma reagin (RPR) test
  * HIV-1 nucleic acid test (NAT)
  * HBV NAT
  * HCV NAT
* Any of the following hematologic abnormalities:

  * Hemoglobin < 9.0 g/dL,
  * ANC < 1,500/μL
  * Platelets < 100,000/μL
* Any of the following serum biochemistry abnormalities:

  * Total bilirubin > 1.5 × ULN
  * AST or ALT > 2.5 × ULN
  * r-GT > 2.5 × ULN
  * ALP > 2.5 × ULN
  * serum albumin < 3.0 g/dL
  * creatinine > 1.5 × ULN
* Female subject who is lactating or has positive serum or urine pregnancy test at Screening Visit
* Female subject with childbearing potential or male subject with female spouse/partner with childbearing potential who refuses to adopt at least two forms of birth control (at least one of which must be a barrier method) from Screening until Final/Early Termination Visit. Acceptable forms include:

  * Established use of oral, injected or implanted hormonal methods of contraception
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * Barrier methods of contraception: condom, or occlusive cap (diaphragm or cervical/vault caps)
* With any condition judged by the investigator that entering the trial may be detrimental to the subject

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Grading of Adverse Events | within 48 weeks after MitoCell transplantation
  Grading will be assessed using NCI CTCAE, version 5.0.
Routine physical examinations | within 48 weeks after MitoCell transplantation
  Safety of Mitocell will be assessed by routine physical examinations. Physical examination conducted in this study will include general appearance, skin, eyes, ears, nose,throat, head and neck, heart, chest and lungs, abdomen, extremities, lymph nodes, musculoskeletal,neurological, etc.
Changes in physical examinations: clinical standard neurological examination [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Clinical standard neurological examination by study investigator. Changes in motor function, sensory function, cranial nerve function (visual fields), cortical functions and reflexes are followed in the examination, scored as normal - abnormal without clinical relevance - abnormal with clinical relevance
Changes in vital signs: blood pressure [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in blood pressure during the study , measured as systolic and diastolic blood pressure (in mmHg)
Changes in vital signs: pulse rate [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in pulse rate during the study (in beats per minute)
Changes in vital signs: body temperature [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in body temperature during the study (in degrees celsius)
Changes in clinical laboratory safety screen: haematology - hemoglobin [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in laboratory variables for haematology: hemoglobin (g/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance"
Changes in clinical laboratory safety screen: Platelet count [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in laboratory variables for haematology: Platelet count (10E9/L). Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance"
Changes in clinical laboratory safety screen: white blood cell (WBC) counts [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in laboratory variables for haematology: Cell counts (10E9/L) for total WBC, neutrophils, lymphocytes, monocytes, eosinophils and basophils. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance"
Changes in clinical laboratory safety screen: International Normalized Ratio (INR) [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in laboratory variables for haematology: INR (standardized prothrombin time) to determine the effects of oral anticoagulants on the clotting system. Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance"
Changes in clinical laboratory safety screen: activated partial thromboplastin time (aPTT) [Safety of Mitocell] | within 48 weeks after MitoCell transplantation
  Changes in laboratory variables for haematology: aPTT (sec) . Result evaluated as "normal", "abnormal without clinical relevance" or "abnormal with clinical relevance"
Electrocardiogram (ECG) | within 48 weeks after MitoCell transplantation
  Safety of Mitocell will be assessed by any clinically significant abnormalities on ECG results as compared to Baseline. A standard 12-lead ECG was measured by using ECG machine that automatically measured PR, QRS, QT, and QTcF intervals.
Magnetic Resonance Imaging (MRI) | within 48 weeks after MitoCell transplantation
  Safety of Mitocell will be assessed by any clinically significant abnormalities on MRI scans as compared to Baseline.

SECONDARY OUTCOMES:
MDS-UPDRS (Movement Disorder Society unified Parkinson's disease rating scale) | at 12, 24, 48 weeks
  Change in MDS-UPDRS motor (Part III) "OFF" score compared to the baseline. All items have 5 response options with uniform anchors of: 0 = normal, 1 = slight (symptoms/signs with sufficiently low frequency or intensity to cause no impact on function), 2 = mild (symptoms/signs of frequency or intensity sufficient to cause a modest impact on function, 3 = moderate (symptoms/signs sufficiently frequent or intense to impact considerably, but not prevent function), 4 = severe (symptoms/signs that prevent function).
Modified Hoehn & Yahr staging | at 12, 24, 48 weeks
  Change in Modified Hoehn & Yahr staging compared to the baseline.
18F-DOPA PET | at 48 weeks
  Degree of radiotracer uptake increment/decrement shown on striatum of 18F-DOPA PET compared to the baseline.
levodopa equivalent daily dose (LEDD) | at 12, 24, 48 weeks
  Reduction of Parkinson's medications consumption by calculating levodopa equivalent daily dose (LEDD) compared to the baseline.
PDQ-39 (Parkinson's Disease Questionnaire) | at 12, 24, 48 weeks
  Change in PDQ-39 scale compared to the baseline. The PDQ-39 is a 39 questions Parkinson's Disease self-completed questionnaire that comprises 8 domains: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). All items are assumed to impact QoL and must be answered to compute scores for each dimension. Questions are answered based on experiences from the preceding month using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.
Beck Depression Inventory (BDI-II) scores | at 48 weeks
  Net change from baseline in BDI-II scores. BDI-II Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
Hamilton Depression Rating Scale (HAM-D-17) scores | at 48 weeks
  Net change from baseline in HAM-D-17 scores. The HAMD-17 is a 17-item assessment used to assess the severity of depression and its improvement during the course of therapy. Each item was evaluated and scored using either a 5-point scale of 0 (not present/absent) to 4 (very severe) or a 3-point scale of 0 (not present/absent) to 2 (marked). Higher scores indicate greater symptom severity. The total score was the sum of the scores from HAMD-17 Items 1 through 17 and ranged from 0 (not at all depressed) to 52 (severely depressed).
Mini Mental State Examination (MMSE) Scores | at 48 weeks
  Net change from baseline in MMSE scores. The MMSE uses a 30 point questionnaire to measure cognitive impairment. The MMSE is scored from 0 to 30,with a score equal to or greater than 24 points indicating normal cognition, a score of 19-23 points indicating mild cognitive impairment, 10-18 points indicating moderate impairment and a score equal to or below 9 indicating severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tang Tu, Ph. D., Study Director — Taiwan Mitochondrion Applied Technology Co., Ltd.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.